CLINICAL TRIAL: NCT05133453
Title: Pirfenidone Use in Asbestosis Patients: Efficacy and Prognosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Mohammed Fouad, Lecturer of Occupational and environmental Medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pirfenidone in asbestosis
Record Dates: First submitted 2021-11-01; First posted 2021-11-24 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Asbestosis
Keywords: Pirfenidone; Asbestosis
MeSH Terms: conditions — Asbestosis | interventions — pirfenidone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pirfinedone group (Active Comparator): asbestosis patients given pirfenidone drug
  Interventions: Drug: Pirfenidone
- Conventional group (No Intervention): Asbestosis patients on conventional treatment

INTERVENTIONS:
Drug: Pirfenidone — drug intake three times daily for one year
  Other Names: Conventional treatment
  Arms: Pirfinedone group

SUMMARY:
This study aims at determining the the efficiency and prognosis of using pirfenidone drug among asbestosis patients.

DETAILED DESCRIPTION:
Asbestos exposure is associated with pleural and lung fibrosis and lung cancer. It has pathomechanisms and clinical similarities to interstitial pulmonary fibrosis disease. There is no definite cure for asbestosis. Pirfenidone has antifibrotic and anti-inflammatory effects.The safety and effectiveness of pirfenidone for the treatment of non-interstitial pulmonary fibrosis progressive fibrotic interstitial lung diseases remain unclear including asbestosis. Only few studies for pirfenidone use in asbestosis.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged ≥ 18 years old
* Patients who fulfilled investigations according the study protocol.
* Patients who kept on follow up for the entire study.
* All patients fulfilling the clinical and radiological criteria of asbestosis (Existence of asbestos-specific pleural changes in high resolution computed topography HRCT (pleural plaques), Reticular changes in HRCT and restrictive lung function pattern, History of asbestos exposure, Absence of an alternative explanation for fibrotic lung disease )
* Clinically stable patients.
* Patients who signed informed consent
* Patients with mild-to-moderate IPF [forced vita capacity (FVC) ≥50% of predicted and diffusion capacity of carbon monoxide (DLCO) ≥30% of predicted].
* Duration since diagnosis (at least one year before the study)

Exclusion Criteria:

* Patients with peptic ulcer,
* Severe hepatic disease, hepatitis C infection or any of the following liver function test criteria above specified limits: aspartate or alanine aminotransferase (AST or ALT) >2.5 u above upper limit of normal level.
* Severe kidney disease, Cardiac disease, and Patients with other chronic pulmonary diseases, lung cancer
* Presence of coexisting respiratory infection
* History of alcohol or drugs abuse
* Patients with neuromuscular disease,
* Chronic renal failure,
* Patient on oxygen therapy,
* Life expectancy less than 6 months,
* History of malignancy.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Ventilatory function change | after 6 months and 12 months from the start of the trial
  Absolute change in percent predicted forced vital capacity
Diffusion test | after 6 months and 12 months from the start of the trial
  Diffusion test change from baseline
radiological findings change | after 6 months and 12 months from the start of the trial
  radiological changes in High resolution computed topography.

CONTACTS AND LOCATIONS:
Overall Officials: Marwa M Fouad, MD, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Behr J, Prasse A, Kreuter M, Johow J, Rabe KF, Bonella F, Bonnet R, Grohe C, Held M, Wilkens H, Hammerl P, Koschel D, Blaas S, Wirtz H, Ficker JH, Neumeister W, Schonfeld N, Claussen M, Kneidinger N, Frankenberger M, Hummler S, Kahn N, Tello S, Freise J, Welte T, Neuser P, Gunther A; RELIEF investigators. Pirfenidone in patients with progressive fibrotic interstitial lung diseases other than idiopathic pulmonary fibrosis (RELIEF): a double-blind, randomised, placebo-controlled, phase 2b trial. Lancet Respir Med. 2021 May;9(5):476-486. doi: 10.1016/S2213-2600(20)30554-3. Epub 2021 Mar 30. PMID 33798455